CLINICAL TRIAL: NCT05368558
Title: A 6-Week, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Cariprazine in the Acute Exacerbation of Schizophrenia, With an Additional 18-Week Blinded Extension Period
Brief Title: Study to Assess Adverse Events and Change in Disease Activity of Oral Cariprazine Capsules in Adult Participants With Schizophrenia
Acronym: 509 JPN Schz
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M22-509
Record Dates: First submitted 2022-05-06; First posted 2022-05-10 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cariprazine; VRAYLAR
MeSH Terms: conditions — Schizophrenia | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cariprazine (Experimental): Participants will receive cariprazine Dose A daily for 6 weeks. Upon completion of 6 week treatment period, participants will have option to receive cariprazine Dose B for 18 weeks.
  Interventions: Drug: Cariprazine
- Placebo (Placebo Comparator): Participants will receive placebo daily for 6 weeks. Upon completion of 6 week treatment period, participants will have option to receive cariprazine Dose B for 18 weeks.
  Interventions: Drug: Cariprazine; Drug: Placebo

INTERVENTIONS:
Drug: Cariprazine — Oral Capsule
  Other Names: VRAYLAR
Drug: Placebo — Oral Capsule
  Arms: Placebo

SUMMARY:
Schizophrenia is a common and severe psychiatric illness characterized by extreme disturbances of cognition and thought, affecting language, perception and sense of self. This study will assess how safe and effective cariprazine is in treating adult participants with schizophrenia in Japan and Taiwan. Adverse events and change in disease activity will be assessed.

Cariprazine (VRAYLAR) is an approved drug for the treatment of schizophrenia in the United States. In the first 6-week period, participants are placed in 1 of 2 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 2 chance that participants will be assigned to placebo. In the next 18-week period, participants will have the option to receive 1 of 3 doses of cariprazine. Approximately 250 adult participants, 18-65 years of age with schizophrenia will be enrolled in approximately 55 sites across Taiwan and Japan.

Participants will receive oral capsules of Cariprazine or placebo for the 6-week Double-blind Period (DBP). Upon completion of 6-week DBP, participants will be eligible to receive oral capsules of Cariprazine for additional 18 weeks in the Blinded Extension Period (BEP), followed by an 8-week safety follow-up period.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

DETAILED DESCRIPTION:
Per the final protocol amendment 3, the number of dosing arms in the 6-week DBP of the study changed from 3 to 2. Participants enrolled in the study through Protocol Amendment 2 and who were randomized to the arm that was eliminated, remained in that arm through DBP and their data are displayed by that arm for the DBP portion of the study in participant flow, baseline characteristics and safety sections. Data for all endpoints are presented as planned per final SAP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with schizophrenia at least 1 year before informed consent.
* Experienced a persistent psychotic episode within 2 months prior to informed consent requiring treatment modifications as judged by the investigator or sub-investigator.

Exclusion Criteria:

- History of clinically significant medical conditions or any other reason that the investigator (or subinvestigator) determines would interfere with the participant's participation in this study or would make the participant an unsuitable candidate to receive study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (52):
- Japan (37):
  - Akita University Hospital /ID# 245941, Akita, Akita
  - International University of Health and Welfare Narita Hospital /ID# 243870, Narita-shi, Chiba
  - Fukuoka University Hospital /ID# 244404, Fukuoka, Fukuoka
  - Kuramitsu Hospital /ID# 242511, Fukuoka, Fukuoka
  - Shiranui Hospital /ID# 243717, Omuta-shi, Fukuoka
  - Gifu University Hospital /ID# 246238, Gifu, Gifu
  - Holy Cross Hospital /ID# 242673, Toki-shi, Gifu
  - Hayakawa Clinic /ID# 242432, Kure, Hiroshima
  - National Hospital Organization Kure Medical Center /ID# 243405, Kure-shi, Hiroshima
  - Goryokai Hospital /ID# 242420, Sapporo, Hokkaido
  - Sapporo Medical University Hospital /ID# 245135, Sapporo, Hokkaido
  - Duplicate_Hokkaido University Hospital /ID# 243245, Sapporo, Hokkaido
  - Kagawa University Hospital /ID# 243772, Kita-gun, Kagawa-ken
  - Taniyama Hospital /ID# 242385, Kagoshima, Kagoshima-ken
  - Yokohama City University Hospital /ID# 244944, Yokohama, Kanagawa
  - Yuge Hospital /ID# 242849, Kumamoto, Kumamoto
  - Duplicate_University Hospital Kyoto Prefectural University of Medicine /ID# 242443, Kyoto, Kyoto
  - Maizuru Medical Center /ID# 243450, Maizuru, Kyoto
  - Mie University Hospital /ID# 244710, Tsu, Mie-ken
  - Mental Support Soyokaze Hospital /ID# 242512, Ueda-shi, Nagano
  - Nara Medical University Hospital /ID# 242561, Kashihara-shi, Nara
  - Asakayama General Hospital /ID# 242732, Sakai, Osaka
  - Hizen Psychiatric Center /ID# 243239, Kanzaki-gun, Saga-ken
  - Rainbow & Sea Hospital /ID# 242699, Karatsu-shi, Saga-ken
  - Inuo Hospital /ID# 243310, Tosu-shi, Saga-ken
  - Juntendo Univ Koshigaya Hospital /ID# 248502, Koshigaya-shi, Saitama
  - Numazu Chuo Hospital /ID# 245275, Numazu-shi, Shizuoka
  - Tochigi Prefectural Okamotodai Hospital /ID# 248855, Utsunomiya, Tochigi
  - Tokushima University Hospital /ID# 250056, Tokushima, Tokushima
  - Narimasu Kosei Hospital /ID# 243107, Banqiao Qu, Tokyo
  - Ongata Hospital /ID# 256975, Hachioji-shi, Tokyo
  - Nishigahara Hospital /ID# 243312, Kita-ku, Tokyo
  - National Center of Neurology and Psychiatry /ID# 242677, Kodaira-shi, Tokyo
  - Tokyo Metropolitan Matsuzawa Hospital /ID# 245272, Setagaya-ku, Tokyo
  - Wakayama Medical University Hospital /ID# 251105, Wakayama, Wakayama
  - Shin-abuyama Hospital /ID# 243138, Takatsuki
  - Minamitoyama Nakagawa Hospital /ID# 243616, Toyama
- Taiwan (15):
  - Kaohsiung Municipal Kai-Syuan Psychiatric Hospital /ID# 241533, Kaohsiung City, Kaohsiung
  - Bali Psychiatric Center /ID# 241597, New Taipei City, New Taipei
  - Taipei Veterans General Hospital /ID# 241522, Taipei City, Taipei
  - Changhua Christian Hospital /ID# 241524, Changhua City, Changhua County
  - National Taiwan University Hospital - Yunlin Branch /ID# 241537, Douliu
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 241528, Kaohsiung City
  - TsaoTun Psychiatric Center, MOHW /ID# 246012, Nantou City
  - New Taipei Municipal TuCheng Hospital (Built and Operated by Chang Gung Medical /ID# 243653, New Taipei City
  - Chung Shan Medical University Hospital /ID# 241543, Taichung
  - Taichung Veterans General Hospital /ID# 246200, Taichung
  - Jianan Psychiatric Center, Ministry of Health and Welfare /ID# 241540, Tainan
  - Taipei City Hospital, Songde Branch /ID# 241600, Taipei
  - Tri-Service General Hospital Beitou Branch /ID# 241563, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 241520, Taoyuan
  - Taoyuan Psychiatric Center, MOHW /ID# 241691, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-509

RESULTS

PARTICIPANT FLOW:
Groups:
- DBP Placebo: Participants received Placebo oral capsule daily for the 6-week Double Blind Period (DBP). Upon completion of 6-week DBP, participants had the option to receive Cariprazine 1.5 mg oral capsule daily for an 18-week Blinded Extension Period (BEP).
- DBP Cariprazine 3 mg: Participants received Cariprazine 3 mg oral capsule daily for the 6-week DBP. Upon completion of 6-week DBP, participants had the option to receive Cariprazine 3 mg oral capsule daily for the 18-week BEP.
- DBP Cariprazine 6 mg: Participants received Cariprazine 6 mg oral capsule daily for the 6-week DBP. Upon completion of 6-week DBP, participants had the option to receive Cariprazine 3 mg oral capsule daily for the 18-week BEP.
- BEP Cariprazine 1.5 mg: Participants who complete the 6-week DBP and moved on to received Cariprazine 1.5 mg modal (most frequent) daily dose during the 18-week BEP.
  Number of participants entered into this arm consisted of:
  N=10 from DBP Placebo
- BEP Cariprazine 3 mg: Participants who complete the 6-week DBP and moved on to received Cariprazine 3 mg modal daily dose during the 18-week BEP.
  Number of participants entered into this arm consisted of:
  N=1 from DBP Placebo N=2 from DBP Cariprazine 3 mg N=1 from DBP Cariprazine 6 mg
- BEP Cariprazine 6 mg: Participants who complete the 6-week DBP and moved on to received Cariprazine 6 mg modal daily dose during the 18-week BEP.
  Number of participants entered into this arm consisted of:
  N=2 from DBP Cariprazine 3 mg N=8 from DBP Cariprazine 6 mg
- SF DBP Placebo: Safety Follow up (SF) for DBP Placebo participants.
- SF DBP Cariprazine 3 mg: SF for DBP Cariprazine 3 mg participants.
- SF DBP Cariprazine 6 mg: SF for DBP Cariprazine 6 mg participants.
- SF BEP Cariprazine 1.5 mg: SF for BEP Cariprazine 1.5 mg participants.
- SF BEP Cariprazine 3 mg: SF for BEP Cariprazine 3 mg participants.
- SF BEP Cariprazine 6 mg: SF for BEP Cariprazine 6 mg participants.
Period: Double Blind Period (DBP)
Arm/Group | DBP Placebo | DBP Cariprazine 3 mg | DBP Cariprazine 6 mg | BEP Cariprazine 1.5 mg | BEP Cariprazine 3 mg | BEP Cariprazine 6 mg | SF DBP Placebo | SF DBP Cariprazine 3 mg | SF DBP Cariprazine 6 mg | SF BEP Cariprazine 1.5 mg | SF BEP Cariprazine 3 mg | SF BEP Cariprazine 6 mg
Started | 16 | 5 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 15 | 4 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Blinded Extension Period (BEP)
Arm/Group | DBP Placebo | DBP Cariprazine 3 mg | DBP Cariprazine 6 mg | BEP Cariprazine 1.5 mg | BEP Cariprazine 3 mg | BEP Cariprazine 6 mg | SF DBP Placebo | SF DBP Cariprazine 3 mg | SF DBP Cariprazine 6 mg | SF BEP Cariprazine 1.5 mg | SF BEP Cariprazine 3 mg | SF BEP Cariprazine 6 mg
Started | 0 | 0 | 0 | 10 | 4 | 10 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 8 | 4 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Safety Follow-up DBP (SF DBP)
Arm/Group | DBP Placebo | DBP Cariprazine 3 mg | DBP Cariprazine 6 mg | BEP Cariprazine 1.5 mg | BEP Cariprazine 3 mg | BEP Cariprazine 6 mg | SF DBP Placebo | SF DBP Cariprazine 3 mg | SF DBP Cariprazine 6 mg | SF BEP Cariprazine 1.5 mg | SF BEP Cariprazine 3 mg | SF BEP Cariprazine 6 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 4 | 11 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 3 | 7 | 0 | 0 | 0
Period: Safety Follow-up BEP (SF BEP)
Arm/Group | DBP Placebo | DBP Cariprazine 3 mg | DBP Cariprazine 6 mg | BEP Cariprazine 1.5 mg | BEP Cariprazine 3 mg | BEP Cariprazine 6 mg | SF DBP Placebo | SF DBP Cariprazine 3 mg | SF DBP Cariprazine 6 mg | SF BEP Cariprazine 1.5 mg | SF BEP Cariprazine 3 mg | SF BEP Cariprazine 6 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 4 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 4 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all randomized participants who received at least 1 dose of study drug.
Groups:
- DBP Placebo: Participants received Placebo oral capsule daily for the 6-week Double Blind Period (DBP). Upon completion of 6week DBP, participants had the option to receive Cariprazine 1.5 mg oral capsule daily for an 18-week Blinded Extension Period (BEP).
- Total: Total of all reporting groups
Arm/Group | DBP Placebo | DBP Cariprazine 3 mg | DBP Cariprazine 6 mg | Total
Number analyzed (Participants) | 16 | 5 | 13 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (11.76) | 40.4 (13.70) | 43.7 (10.88) | 42.5 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 6 | 13
  Male | 10 | 4 | 7 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 5 | 13 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 16 | 5 | 13 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
SCI-PANSS Total Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — Structured Clinical Interview for the Positive and Negative Syndrome Scale (SCI-PANSS) is a 30-item clinician-reported rating scale which assesses both the positive and negative symptom syndromes of patients with schizophrenia. This assessment provides scores in 9 clinical domains, including a positive syndrome, a negative syndrome, depression, a composite index, and general psychopathology. Each item is scored on a 7-point scale with responses ranging from 1 (absent) to 7 (extreme). The SCI-PANSS total score can range from 30 to 210. Higher values represent a worse outcome.
  score on a scale | 94.6 (8.70) | 99.8 (8.17) | 91.8 (7.37) | 94.3 (8.33)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Time Frame: From first dose of study drug until 8 weeks following last dose of study drug (up to 32 weeks)
Population: Safety Population includes all randomized participants who receive at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DBP Placebo | DBP Cariprazine 3 mg | DBP Cariprazine 6 mg
Number analyzed (Participants) | 16 | 5 | 13
Participants | 12 | 2 | 10

2. Primary Outcome: Change in SCI-PANSS Total Score From Baseline (Wk 0) to Week 6.
Description: Structured Clinical Interview for the Positive and Negative Syndrome Scale (SCI-PANSS) is a 30-item clinician-reported rating scale which assesses both the positive and negative symptom syndromes of patients with schizophrenia. This assessment provides scores in 9 clinical domains, including a positive syndrome, a negative syndrome, depression, a composite index, and general psychopathology. Each item is scored on a 7-point scale with responses ranging from 1 (absent) to 7 (extreme). Higher values represent a worse outcome. The SCI-PANSS total score can range from 30 to 210. A negative change from baseline indicates improvement.
Time Frame: Baseline (Wk 0) to Week 6
Population: mITT Population includes all randomized participants who receive at least 1 dose of study drug and have both baseline and at least 1 postbaseline value during the DBP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBP Placebo | DBP Cariprazine 3 mg | DBP Cariprazine 6 mg
Number analyzed (Participants) | 11 | 5 | 10
score on a scale | -15.2 (12.21) | -5.6 (10.38) | -30.2 (17.47)
Statistical Analysis 1: Comparison: DBP Placebo vs DBP Cariprazine 3 mg; Test type: Superiority; Mean Difference (Final Values) = 9.6, 95% CI 2-sided [-4.0 to 23.1]
Statistical Analysis 2: Comparison: DBP Placebo vs DBP Cariprazine 6 mg; Test type: Superiority; Mean Difference (Final Values) = -15.0, 95% CI 2-sided [-28.7 to -1.4]

3. Secondary Outcome: Change in CGI-S Score From Baseline (Wk 0) to Week 6
Description: Clinical Global Impression-Severity (CGI-S) is a single, clinician-reported item that measures the clinician's impression of a participant's current anxiety severity considering their total clinical experience with the patient population. The measure uses a 7-point Likert rating scale with responses ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The total CGI-S score can range from 1 to 7. A higher score indicates more severe illness. A negative change from baseline indicates improvement.
Time Frame: Baseline (Wk 0) to Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBP Placebo | DBP Cariprazine 3 mg | DBP Cariprazine 6 mg
Number analyzed (Participants) | 11 | 5 | 10
score on a scale | -0.6 (0.92) | -0.4 (0.55) | -1.3 (1.25)
Statistical Analysis 1: Comparison: DBP Placebo vs DBP Cariprazine 3 mg; Test type: Superiority; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.7 to 1.2]
Statistical Analysis 2: Comparison: DBP Placebo vs DBP Cariprazine 6 mg; Test type: Superiority; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.7 to 0.3]

4. Secondary Outcome: Change in SCI-PANSS Positive Symptom Score From Baseline (Wk 0) to Week 6
Description: as for outcome 2
Time Frame: Baseline (Wk 0) to Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBP Placebo | DBP Cariprazine 3 mg | DBP Cariprazine 6 mg
Number analyzed (Participants) | 11 | 5 | 10
score on a scale | -4.7 (4.67) | -2.2 (3.35) | -8.7 (4.00)
Statistical Analysis 1: Comparison: DBP Placebo vs DBP Cariprazine 3 mg; Test type: Superiority; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-2.5 to 7.5]
Statistical Analysis 2: Comparison: DBP Placebo vs DBP Cariprazine 6 mg; Test type: Superiority; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-8.0 to 0.0]

5. Secondary Outcome: Change in NSA-16 Total Score to Baseline (Wk 0) to Week 6
Description: Negative Symptom Assessment-16 (NSA-16) is a 16-item clinician-reported scale covering 5 areas or domains: communication, affect, social involvement, motivation, and retardation. It is designed to assess negative symptoms of patients with schizophrenia. Each item or behavior is rated on a 6-point scale ranging from 1 (not reduced) to 6 (severely reduced or absent). Higher values represent a worse outcome. The total NSA-16 score can range from 16 to 96. A negative change from baseline indicates improvement.
Time Frame: Baseline (Wk 0) to Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBP Placebo | DBP Cariprazine 3 mg | DBP Cariprazine 6 mg
Number analyzed (Participants) | 11 | 5 | 10
score on a scale | -3.2 (7.49) | -2.8 (9.20) | -14.5 (8.28)
Statistical Analysis 1: Comparison: DBP Placebo vs DBP Cariprazine 3 mg; Test type: Superiority; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-8.9 to 9.7]
Statistical Analysis 2: Comparison: DBP Placebo vs DBP Cariprazine 6 mg; Test type: Superiority; Mean Difference (Final Values) = -11.3, 95% CI 2-sided [-18.5 to -4.1]

6. Secondary Outcome: Change in SCI-PANSS Negative Symptom Score From Baseline (Wk 0) to Week 6
Description: as for outcome 2
Time Frame: Baseline (Wk 0) to Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBP Placebo | DBP Cariprazine 3 mg | DBP Cariprazine 6 mg
Number analyzed (Participants) | 11 | 5 | 10
score on a scale | -3.5 (3.86) | -0.2 (3.27) | -8.1 (5.30)
Statistical Analysis 1: Comparison: DBP Placebo vs DBP Cariprazine 3 mg; Test type: Superiority; Mean Difference (Final Values) = 3.3, 95% CI 2-sided [-1.0 to 7.5]
Statistical Analysis 2: Comparison: DBP Placebo vs DBP Cariprazine 6 mg; Test type: Superiority; Mean Difference (Final Values) = -4.6, 95% CI 2-sided [-8.9 to -0.4]

7. Secondary Outcome: Change in SCI-PANSS Negative Factor Score From Baseline (Wk 0) to Week 6
Description: as for outcome 2
Time Frame: Baseline (Wk 0) to Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBP Placebo | DBP Cariprazine 3 mg | DBP Cariprazine 6 mg
Number analyzed (Participants) | 11 | 5 | 10
score on a scale | -3.8 (3.71) | -0.4 (3.78) | -9.1 (6.82)
Statistical Analysis 1: Comparison: DBP Placebo vs DBP Cariprazine 3 mg; Test type: Superiority; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [-0.9 to 7.7]
Statistical Analysis 2: Comparison: DBP Placebo vs DBP Cariprazine 6 mg; Test type: Superiority; Mean Difference (Final Values) = -5.3, 95% CI 2-sided [-10.2 to -0.3]

8. Secondary Outcome: Change in SCI-PANSS Total Score From Baseline (Wk 0) and Week 6 to Week 24
Description: as for outcome 2
Time Frame: Baseline (Wk 0) and Week 6 to Week 24
Population: BEP population consisted of all participants who complete the 6-week DBP and received at least 1 dose of study drug during the BEP regardless of which treatment group they were randomized to during the DBP.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BEP Cariprazine 1.5 mg: Participants who complete the 6-week DBP and moved on to received Cariprazine 1.5 mg modal (most frequent) daily dose during the 18-week BEP.
- BEP Cariprazine 3 mg: Participants who complete the 6-week DBP and moved on to received Cariprazine 3 mg modal daily dose during the 18-week BEP.
- BEP Cariprazine 6 mg: Participants who complete the 6-week DBP and moved on to received Cariprazine 6 mg modal modal daily dose during the 18-week BEP.
Arm/Group | BEP Cariprazine 1.5 mg | BEP Cariprazine 3 mg | BEP Cariprazine 6 mg
Number analyzed (Participants) | 5 | 3 | 4
score on a scale
  Baseline (Wk 0) to Week 24 | -19.2 (19.52) | -19.3 (30.09) | -22.5 (25.16)
  Week 6 to Week 24 | -4.0 (16.05) | 2.0 (4.58) | 6.0 (17.51)

9. Secondary Outcome: Change in CGI-S Score From Baseline (Wk 0) and Week 6 to Week 24
Description: as for outcome 3
Time Frame: Baseline (Wk 0) and Week 6 to Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BEP Cariprazine 1.5 mg | BEP Cariprazine 3 mg | BEP Cariprazine 6 mg
Number analyzed (Participants) | 5 | 3 | 4
score on a scale
  Baseline (Wk 0) to Week 24 | -0.8 (0.84) | -1.3 (2.31) | -1.0 (0.82)
  Week 6 to Week 24 | -0.4 (1.14) | 0.0 (0.00) | 0.0 (0.82)

10. Secondary Outcome: Change in SCI-PANSS Positive Symptom Score From Baseline (Wk 0) and Week 6 to Week 24
Description: as for outcome 2
Time Frame: Baseline (Wk 0) and Week 6 to Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BEP Cariprazine 1.5 mg | BEP Cariprazine 3 mg | BEP Cariprazine 6 mg
Number analyzed (Participants) | 5 | 3 | 4
score on a scale
  Baseline (Wk 0) to Week 24 | -5.2 (5.36) | -4.3 (7.51) | -6.8 (6.60)
  Week 6 to Week 24 | -0.2 (4.38) | 0.3 (0.58) | 1.5 (6.03)

11. Secondary Outcome: Change in NSA-16 Total Score From Baseline (Wk 0) and Week 6 to Week 24
Description: as for outcome 5
Time Frame: Baseline (Wk 0) and Week 6 to Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BEP Cariprazine 1.5 mg | BEP Cariprazine 3 mg | BEP Cariprazine 6 mg
Number analyzed (Participants) | 5 | 3 | 4
score on a scale
  Baseline (Wk 0) to Week 24 | -11.6 (13.52) | -5.0 (14.00) | -13.3 (20.19)
  Week 6 to Week 24 | -7.6 (18.28) | 2.7 (5.51) | -1.8 (11.18)

12. Secondary Outcome: Change in SCI-PANSS Negative Symptom Score From Baseline (Wk 0) and Week 6 to Week 24
Description: as for outcome 2
Time Frame: Baseline (Wk 0) and Week 6 to Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BEP Cariprazine 1.5 mg | BEP Cariprazine 3 mg | BEP Cariprazine 6 mg
Number analyzed (Participants) | 5 | 3 | 4
score on a scale
  Baseline (Wk 0) to Week 24 | -6.4 (3.85) | -5.0 (6.24) | -5.3 (9.64)
  Week 6 to Week 24 | -2.8 (4.09) | -1.3 (2.52) | 2.3 (4.19)

13. Secondary Outcome: Change in SCI-PANSS Negative Factor Score From Baseline (Wk 0) and Week 6 to Week 24
Description: as for outcome 2
Time Frame: Baseline (Wk 0) and Week 6 to Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BEP Cariprazine 1.5 mg | BEP Cariprazine 3 mg | BEP Cariprazine 6 mg
Number analyzed (Participants) | 5 | 3 | 4
score on a scale
  Baseline (Wk 0) to Week 24 | -5.2 (4.09) | -6.7 (9.29) | -6.0 (9.76)
  Week 6 to Week 24 | -1.6 (3.78) | -1.0 (1.00) | 2.0 (4.16)

ADVERSE EVENTS:
Time Frame: All-cause mortality were reported from enrollment to the end of study. In the DBP, median time on follow up (median time subjects were followed) was 42.0 days (d) for all arms (DBP: Pbo, C 3mg, and C 6mg). In the BEP, median time on follow up was 117.5, 126.0, and 97.5d for BEP: C1.5mg, C 3mg, and C 6mg, respectively. In the SF DBP, median time on follow up was 57.0, 1.0, and 47.0d for SF DBP: Pbo, C 3mg, and C 6mg, respectively.
Description: In the SF BEP, median time on follow up was 56.0, 57.0, and 56.5d for SF BEP: C1.5mg, C 3mg, and C 6mg, respectively. Treatment-emergent adverse events and serious adverse events were collected from first dose of study drug until 8 weeks after the last dose of study drug. Mean duration on study drug was 36.4, 41.8, and 38.9d for DBP: Pbo, C 3mg, and C 6mg, respectively. Mean duration on study drug was 88.2,108.5, and 87.1d for BEP: C1.5mg, C 3mg, and C 6mg, respectively.
Groups:
- BEP Cariprazine 1.5 mg: Participants who complete the 6-week DBP and moved on to received Cariprazine 1.5 mg modal modal (most frequent) daily dose during the 18-week BEP.
- BEP Cariprazine 3 mg: Participants who complete the 6-week DBP and moved on to received Cariprazine 3 mg modal modal (most frequent) daily dose during the 18-week BEP.
- BEP Cariprazine 6 mg: Participants who complete the 6-week DBP and moved on to received Cariprazine 6 mg modal modal (most frequent) daily dose during the 18-week BEP.
Arm/Group | DBP Placebo | DBP Cariprazine 3 mg | DBP Cariprazine 6 mg | BEP Cariprazine 1.5 mg | BEP Cariprazine 3 mg | BEP Cariprazine 6 mg | SF DBP Placebo | SF DBP Cariprazine 3 mg | SF DBP Cariprazine 6 mg | SF BEP Cariprazine 1.5 mg | SF BEP Cariprazine 3 mg | SF BEP Cariprazine 6 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/5 | 0/13 | 0/10 | 0/4 | 0/10 | 0/5 | 0/1 | 0/4 | 0/10 | 0/4 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/5 | 0/13 | 1/10 | 1/4 | 0/10 | 0/5 | 0/1 | 1/4 | 0/10 | 1/4 | 0/10
Other Adverse Events (participants affected / at risk) | 12/16 | 2/5 | 10/13 | 7/10 | 3/4 | 6/10 | 3/5 | 0/1 | 2/4 | 4/10 | 0/4 | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBP Placebo (N=16) | DBP Cariprazine 3 mg (N=5) | DBP Cariprazine 6 mg (N=13) | BEP Cariprazine 1.5 mg (N=10) | BEP Cariprazine 3 mg (N=4) | BEP Cariprazine 6 mg (N=10) | SF DBP Placebo (N=5) | SF DBP Cariprazine 3 mg (N=1) | SF DBP Cariprazine 6 mg (N=4) | SF BEP Cariprazine 1.5 mg (N=10) | SF BEP Cariprazine 3 mg (N=4) | SF BEP Cariprazine 6 mg (N=10)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SCHIZOPHRENIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBP Placebo (N=16) | DBP Cariprazine 3 mg (N=5) | DBP Cariprazine 6 mg (N=13) | BEP Cariprazine 1.5 mg (N=10) | BEP Cariprazine 3 mg (N=4) | BEP Cariprazine 6 mg (N=10) | SF DBP Placebo (N=5) | SF DBP Cariprazine 3 mg (N=1) | SF DBP Cariprazine 6 mg (N=4) | SF BEP Cariprazine 1.5 mg (N=10) | SF BEP Cariprazine 3 mg (N=4) | SF BEP Cariprazine 6 mg (N=10)
DRY EYE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IRIDOCYCLITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UVEITIS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DENTAL CARIES (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEELING ABNORMAL (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HORDEOLUM (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIODONTITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHILLBLAINS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IMMUNISATION REACTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST VACCINATION SYNDROME (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WOUND (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CHLORIDE DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD SODIUM DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HIGH DENSITY LIPOPROTEIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WEIGHT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AKATHISIA (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PARKINSONISM (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOGORRHOEA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NIGHTMARE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESTLESSNESS (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SCHIZOPHRENIA (Psychiatric disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSMENORRHOEA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SCROTAL ERYTHEMA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT05368558/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT05368558/SAP_001.pdf